CLINICAL TRIAL: NCT03364439
Title: Prospective, Multicentre Phase II Study With R-CHOP- 14 or R-CHOP-21 & Consolidation PET-Oriented Radiotherapy (RT) in Diffuse Large B Cell Lymphoma (DLBCL) Patients With Low Risk Profile According to Age-adjusted IPI (0 With Bulky or 1)
Brief Title: R-CHOP14 or R-CHOP21 &Consolidation PET-Oriented Radiotherapy (RT) in DLBCL Patients
Acronym: FIL_DLCL10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_DLCL10
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm for all patients (Experimental): Patients eligible for the study will receive 6 courses of R-CHOP14 or R-CHOP21.
  Interventions: Drug: Treatment plan

INTERVENTIONS:
Drug: Treatment plan — R-CHOP14 or R-CHOP21 for 6 cycles Restaging after 2, 4, 6 cycles Consolidation therapy with RT (36 Gy) if PET positive (PET after 6 R-CHOP cycles)

SUMMARY:
Prospective, multicentre phase II study with R-CHOP- 14 or R-CHOP-21 & consolidation PET-oriented radiotherapy (RT) in diffuse large B cell lymphoma (DLBCL) patients

DETAILED DESCRIPTION:
Prospective, multicentre phase II study with R-CHOP- 14 or R-CHOP-21 & consolidation PET-oriented radiotherapy (RT) in diffuse large B cell lymphoma (DLBCL) patients with low risk profile according to age-adjusted IPI (0 with bulky or 1)

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of DLBCL (CD20+), follicular lymphoma grade IIIB, T-cell rich large B cell lymphoma
* Age 18-80 years (patients >70 years old: FIT according to VGM evaluation).
* aaIPI=1 +/- bulky and aaIPI=0 with bulky (>7.5 cm)
* ECOG-PS < 3 unless due to lymphoma
* Ventricular ejection fraction ≥ 50%
* Pulmonary, renal and hepatic tests within normal range
* Negative HIV and HBV tests. In case of HBcAb positive and HBsAb +/-, which is indicative of a past infection (occult carriers) the subject can be included, but antiviral prophylaxis with lamivudine must be given from the beginning of treatment until 12 months after treatment completion. Anti-HCV positive patients can be included in the absence of viral replication (HVR-RNA absent or less than 500 copies/ml.
* Written informed consent
* Life-expectancy > 3 months

Main Exclusion Criteria:

* T-cell lymphoma
* Follicular lymphoma (grade I, II, IIIA), marginal zone and mantle lymphoma
* PS> 3 (if not due to lymphoma)
* Age-adjusted IPI = 0 in the absence of bulky disease
* Age> 80 and <18 years (see inclusion criteria)
* HIV positivity
* significant cardiopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-01; Primary Completion 2018-04 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
PFS Progression Free Survival | 24 months
  defined as non response after 4 or 6 cycles of chemotherapy or progression of disease after consolidation RT or at any time of therapy, relapse or death from any cause.

SECONDARY OUTCOMES:
OS Overall Survival | 48 months
  OS will be defined as the time between the date of initiation of therapy and the date of death from any cause or the date of last follow up

CONTACTS AND LOCATIONS:
Overall Officials: Maria Giuseppina Cabras, Principal Investigator — Ospedale Businco di Cagliari
Locations (19):
- Italy (19):
  - A.O. Niguarda, Milan, MI
  - Centro di Riferimento Oncologico della Basilicata, Rionero in Vulture, PZ
  - A.O. SS. Antonio e Biagio e C. Arrigo, Alessandria
  - A.O. Universitaria Ospedali Riuniti - Ospedale Umberto I Di Ancona, Ancona
  - Centro di riferimento Oncologico Oncologia Medica A, Aviano
  - Ospedale Degli Infermi - S.C. Oncologia, Biella
  - A.O. Spedali Civili di Brescia - Ematologia, Brescia
  - PO Perrino, Brindisi
  - Ospedale Businco, Cagliari
  - Ospedale di Castelfranco Veneto - Ematologia, Castelfranco Veneto
  - Osp.Generale Di Zona Valduce, Como
  - Osp. San Carlo Borromeo Divisione di Oncologia Medica, Milan
  - A.O. Universitaria Maggiore Della Carita' Di Novara, Novara
  - AOU di Parma UO Ematologia e CTMO, Parma
  - Ausl Di Piacenza, Piacenza
  - AO Arcispedale S.Maria Nuova Ematologia, Reggio Emilia
  - Istituto Clinica Humanitas, Rozzano (MI)
  - A.O.U. Citta della Salute e della Scienza di Torino - SC Ematologia, Torino
  - A.O.U. Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino